CLINICAL TRIAL: NCT07340021
Title: Effects of Neuromuscular Warm-up Versus Conventional Warm-up Protocols on Dynamic Balance and Strength Among Recreational Gym Population
Brief Title: Comparative Study of Effects of Neuromuscular Warmup vs Conventional Warmup in Recreational Gym Population
Acronym: NMWU YBT CMJ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lahore University of Biological and Applied Sciences (Other)
Responsible Party: Principal Investigator, Prof. Dr. Shoaib Waqas, Prof. Dr. Shoaib Waqas, Lahore University of Biological and Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: DPT/ERB/42; U1111-1333-1918 (Registry Identifier: Muhammad Ibrahim)
Record Dates: First submitted 2026-01-05; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Participants; Gym Population is Being Studied to Enhance Their Balance and Strength for Better Injury Prevention
Keywords: Gym-Goers; Neuromuscular Warm-up; Conventional Warm-up; Dynamic Balance; Strength; Recreational Gym Population

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neuromuscular Warm-up (Experimental): Participants in the experimental group performed a neuromuscular warm-up program, prior to their training , designed to improve dynamic balance, strength via YBT and vertical jump along with overall neuromuscular control before their regular gym workouts. This warm-up focused on coordinated, functional movements that challenge postural stability and promote efficient muscle activation. The program included progressive balance tasks, controlled strength exercises, agility drills, and dynamic stability activities aimed at activating the neuromuscular system in a purposeful manner. slight progression was made every week All sessions were supervised to ensure correct technique, appropriate progression and the participant safety throughout the intervention period
  Interventions: Behavioral: NM Warm-up
- Conventional Warm-up (Active Comparator): Participants in the control group performed a traditional warm-up routine that was different from the neuromuscular warm-up used in the experimental group. This approach mainly focused on getting the body ready for exercise by increasing heart rate and loosening the muscles, rather than improving neuromuscular control. Unlike the neuromuscular warm-up, this protocol did not include balance-challenging exercises, reactive movements, or tasks that required high levels of body awareness. The movements were simple and repetitive, with no added progression in difficulty, and were intended only to prepare participants physically before starting their regular gym workout.
  Interventions: Behavioral: Conventional Warm-up

INTERVENTIONS:
Behavioral: NM Warm-up — The neuromuscular warm-up was performed four times per week for six weeks, with each session lasting approximately 10 to12 minutes at light to moderate intensity. The intervention consisted of single-leg balance exercises with reach tasks, bosu mini squats with controlled tempo, core stabilization exercises such as front and side planks, and agility-based movements including lateral shuffles and hops. Exercise difficulty was progressively increased by altering base of support, movement speed, and task complexity. The sequence was designed to improve motor control, balance reactions, and force production before the main workout. Dynamic balance and strength outcomes were assessed at baseline and after completion of the intervention.
  Arms: Neuromuscular Warm-up
Behavioral: Conventional Warm-up — Participants in the control group completed the conventional warm-up four times per week for six weeks, with each session lasting about 10 to 12 minutes. The warm-up began with light aerobic activity, such as treadmill jogging or stationary cycling, to gently raise heart rate and body temperature. This was followed by dynamic mobility and stretching exercises, including leg swings, arm circles, hip rotations, , body-weight squats, and dynamic stretches for the hamstrings and calves also of upper body dynamic stretches . Overall, the conventional warm-up aimed to prepare the muscles and joints for exercise but did not specifically target neuromuscular activation, balance, or movement control.
  Arms: Conventional Warm-up

SUMMARY:
* Impaired balance or insufficient strength may increase the risk of musculoskeletal injuries among recreational enthusiasts. Warm-up protocols are an essential component of exercise preparation, aiming to enhance performance and reduce the risk of injury among physically active individuals.
* Neuromuscular warm-up protocols are designed to stimulate the sensorimotor system by integrating balance, coordination, strength, and proprioceptive exercises. These protocols enhance neuromuscular control, joint stability, and muscle activation, which are critical for dynamic movements performed during gym-based training and functional activities.
* Similarly, Conventional warm-up protocols consist of light aerobic activity and static or dynamic stretching. These protocols enhance blood flow and muscle flexibility.
* Dynamic balance refers to the ability to maintain postural control while performing movement tasks and is a key determinant of athletic performance and injury prevention.
* Strength is an essential component for functional performance and is commonly assessed through Counter jump movement tests.
* This study aims to compare the effects of a neuromuscular warm-up versus a conventional warm-up on dynamic balance and strength among recreational gym enthusiasts. The findings may help create a more effective warm-up strategy for improving performance in recreational enthusiasts.

DETAILED DESCRIPTION:
Experimental Group (Neuromuscular Warm-up Protocol):

Participants assigned to the experimental group underwent a structured neuromuscular warm-up (NM-W) program before their routine gym training sessions. The intervention was conducted four times per week over a period of six weeks, with each warm-up session lasting approximately 10-12 minutes at a low to moderate intensity. The protocol began with a light aerobic phase, consisting of treadmill jogging at 50-60% of maximum heart rate for two minutes, followed by dynamic mobility exercises such as arm circles and leg swings. This was followed by a core activation and strengthening phase, which included front planks, side planks, and single-leg glute bridges aimed at enhancing trunk stability and proximal muscle control. The final phase focused on balance and plyometric activities, including single-leg balance with eyes closed, step-ups, BOSU mini squats, and diagonal hopping drills combined with medicine-ball interception gestures. This neuromuscular warm-up protocol was specifically designed to improve neuromuscular integration, enhance dynamic balance, and increase muscular strength prior to resistance-based training.

Control Group ( conventional warmup Protocol):

Participants allocated to the control group received a conventional (traditional) warm-up protocol prior to their routine workout sessions. The warm-up was performed four times per week for six weeks same as in experimental group, with each session lasting approximately 12 minutes, matching the frequency and duration of the experimental group. The conventional warm-up consisted of a general aerobic component aimed at increasing body temperature and heart rate, followed by dynamic mobility exercises. The aerobic phase included treadmill jogging at 50-60% of maximum heart rate for approximately five minutes, after which participants performed dynamic movements such as leg swings, dynamic hip circles, arm swings, high knees, and butt kicks. The overall intensity of the warm-up was maintained at a low to moderate level (RPE 4-5). This protocol was intended to enhance blood circulation, improve muscle flexibility, and prepare the musculoskeletal system for subsequent exercise, without targeting specific neuromuscular, balance, or plyometric training components.

ELIGIBILITY:
Inclusion Criteria:

* Adults age ranging from 18 to 40 years
* No injury at the start of the study
* Willingness to attend all warmup sessions for 6 weeks
* Recreationally Active individuals who participates in exercise for ≥4 times per week
* Individuals who take part in Strength based training and perform closed kinematic chain exercises at least 2 times per week

Exclusion Criteria:

* Any known cardiovascular, systemic illness that might hinder exercises
* History of any injury or surgery in the past 6 months
* Diagnosed neurological, musculoskeletal disorders
* Participation in any competitive professional sports or athletic training

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Dynamic Balance | 8 weeks
  Dynamic balance will be measured using the Y-Balance Test (YBT).
  The Y-Balance Test assesses dynamic postural control by measuring reach distance in three directions while maintaining single-leg stance. The test has demonstrated good to excellent reliability with an internal consistency of Cronbach's alpha (α) of approximately 0.91.
  Y-Balance Test Directions:
  1. Anterior Reach: ______ cm
  2. Posteromedial Reach: ______ cm
  3. Posterolateral Reach: ______ cm Composite Y-Balance Score: ______ % The composite score will be calculated by normalizing reach distances to limb length.
Strength | 8 weeks
  Lower limb strength will be measured using the Countermovement Jump (CMJ) Test. The CMJ test evaluates explosive lower extremity strength by measuring vertical jump height. The MyJump2 smartphone application has demonstrated excellent internal consistency, with a reported Cronbach's alpha (α) of approximately 0.99,This indicates high level of reliability for measuring counter movement jump(CMJ height)
  Countermovement Jump Variables:
  Jump Height: ______ cm

CONTACTS AND LOCATIONS:
Overall Officials: Shoaib Waqas, Phd, Study Chair — Lahore University of Biological and Applied Sciences; Muhammad Ibrahim, DPT, Principal Investigator — Lahore College of Physical Therapy; Muhammad Zoraiz Khan, DPT, Principal Investigator — Lahore College of Physical Therapy; Dua Ali Memon, DPT, Principal Investigator — Lahore College of Physical Therapy
Locations (1):
- Lahore University of Biological and Applied Sciences, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
After the Publication
Supporting Information: Study Protocol, SAP
Time Frame: June 2026- October 2026